CLINICAL TRIAL: NCT03721263
Title: A Phase 1, Open-Label, Single Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of ASLAN004 in Healthy Subjects
Brief Title: Study of ASLAN004 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ASLAN Pharmaceuticals (Other)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASLAN004-001
Record Dates: First submitted 2018-10-10; First posted 2018-10-26 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Allergic Disorder
Keywords: Allergic disorder
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Single Ascending Dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASLAN004 Single Ascending Dose (Experimental): Up to 10 dose levels are planned.
  ASLAN004 by IV route: 0.1 mg/kg (Cohort 1), 0.3 mg/kg (Cohort 2), 1 mg/kg (Cohort 3), 3 mg/kg (Cohort 4) and 10 mg/kg (Cohort 5), 20 mg/kg (Cohort 6 [optional]).
  ASLAN004 SC route: 75 mg (Cohort 7), 150 mg (Cohort 8), 300 mg (Cohort 9), and 600 mg (Cohort 10 [optional]).
  Interventions: Biological: ASLAN004

INTERVENTIONS:
Biological: ASLAN004 — Single Dose

SUMMARY:
This is an open-label, two-part, single-center, first in human (FIH), single ascending dose (SAD) study to assess the effects of single doses of ASLAN004 when administered to healthy subjects. The objective of this study is to evaluate the safety, tolerability, and Pharmacokinetics (PK) of ASLAN004 in healthy subjects.

DETAILED DESCRIPTION:
The plan is to enroll between 38 to 50 subjects at 1 study center.

The study is divided into 2 parts:

Part A is designed as a SAD study using intravenous (IV) administration of ASLAN004, as a single mg/kg IV dose and will consist of up to 6 IV cohorts.

Part B is designed as a parallel SAD study using subcutaneous (SC) administration of ASLAN004, as a single fixed milligram SC dose and will consist of up to 4 SC cohorts.

All cohorts will have sentinel dosing with the first subject of each cohort being spaced with adequate observation time of 24 to 48 hours before dosing the remaining subjects in the cohort.

All subjects would be follow up for up to 85 days from the last dosing day.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to sign informed consent form
2. Male and female subjects who are of legal age
3. Healthy, BMI 18.5 to 30 kg/m2
4. Normal or clinically acceptable clinical laboratory value and ECG results

Exclusion Criteria:

1. History of hypersensitivity reaction
2. Have food and/or topical allergies
3. Have recent history of conjunctivitis
4. Have active or history of psoriasis

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of product safety by assessing the incidence of treatment-emergent adverse events following single ascending dose administration in healthy volunteers at Day 1 until study completion | 85 days
  To evaluate the safety of the product by assessing its impact on the healthy volunteer following single dose administration through review of adverse event listings

SECONDARY OUTCOMES:
PK parameters: Area under the curve (AUC) from time zero to the time of the last quantifiable concentration [AUC(0-last)] | Predose,1 hour, 2 hour, 4 hour, 8 hour, 24 hour, 72 hour, 168 hour, 240 hour and up to 3 months
  To assess the pharmacokinetics of ASLAN004 in healthy volunteers following single dose administration via IV or SC route (16 timepoints)
PK parameters: Estimate of volume of distribution at steady state (Vss) | Predose,1 hour, 2 hour, 4 hour, 8 hour, 24 hour, 72 hour, 168 hour, 240 hour and up to 3 months
  To assess the pharmacokinetics of ASLAN004 in healthy volunteers following single dose administration via IV or SC route (16 timepoints)
PK parameters: Subcutaneous bioavailability (F) | Predose,1 hour, 2 hour, 4 hour, 8 hour, 24 hour, 72 hour, 168 hour, 240 hour and up to 3 months
  To assess the pharmacokinetics of ASLAN004 in healthy volunteers following single dose administration via SC route only (16 timepoints)
PK parameters: Dose-normalized Cmax (Cmax/dose) | Predose,1 hour, 2 hour, 4 hour, 8 hour, 24 hour, 72 hour, 168 hour, 240 hour and up to 3 months
  To assess the pharmacokinetics of ASLAN004 in healthy volunteers following single dose administration via IV or SC route (16 timepoints)
PK parameters: AUC (AUC(0-inf)/dose) | Predose,1 hour, 2 hour, 4 hour, 8 hour, 24 hour, 72 hour, 168 hour, 240 hour and up to 3 months
  To assess the pharmacokinetics of ASLAN004 in healthy volunteers following single dose administration via IV or SC route (16 timepoints)

CONTACTS AND LOCATIONS:
Locations (1):
- CGH Clinical Trials & Research Unit, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No